CLINICAL TRIAL: NCT02869893
Title: Magnetic Resonance Cholangiopancreatography (MRCP): A Reliable, Non Invasive Method for Staging Chronic Pancreatitis From Minimal Change Disease to the Advanced Stages in Pediatrics
Brief Title: MRCP: A Reliable, Non Invasive Method for Staging Chronic Pancreatitis in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: ChiRhoClin, Inc. (Industry); The National Pancreas Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIN_MRCPStudy_001
Record Dates: First submitted 2016-06-05; First posted 2016-08-17 (Estimated); Results first posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Secretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Participants (Other): MRCP with Secretin and MR elastography will be performed on all participants.
  Interventions: Drug: Secretin

INTERVENTIONS:
Drug: Secretin
  Other Names: ChiRhoStim

SUMMARY:
The goal of this research study is to learn more about the pancreas. The investigators want to use Magnetic Resonance Cholangiopancreatography (MRCP) to learn more about the size of a normal pancreas. MRCP is a special kind of MRI exam that produces detailed images of the pancreas. The investigators also want to figure out how much fluid the pancreas releases in response to secretin. Secretin is a chemical in the body that causes the pancreas to release fluid that helps with digestion. Secretin is used during the MRCP (MR-PFT) to help identify dysfunction of the pancreas. MR elastography (MRE) will be used to measure how hard the pancreas is. MRE is a special kind of MRI that uses vibrations to image tissue.

DETAILED DESCRIPTION:
Introduction/Methods: Pancreatic fibrosis is the end stage of chronic pancreatitis (CP), which leads to loss of acinar volume and secretory capacity, and ultimately pancreatic insufficiency (PI). CP and congenital PI affect the pediatric population, and are both increasingly recognized in children. PI has serious negative implications on a child's growth and health but, if diagnosed early, PI can be treated, minimizing the detrimental effects of PI. Currently, direct pancreatic function testing (PFT) via collection of pancreatic fluid is the "gold standard" for diagnosis of PI but it is an invasive testing that may require sedation or general anesthesia. Magnetic resonance cholangiopancreatography (MRCP) with secretin administration (MR-PFT) and MR elastography (MRE) may allow non-invasive, and potentially early diagnosis of CP and PI. Currently, however, normative data with which to compare MR-PFT and MRE results in pediatric patients with suspected CP/PI is not available.

Aims: The investigators propose to determine the normal range for secreted pancreatic fluid volume in response to secretin administration and determine the normal range for pancreatic parenchymal stiffness in a pediatric population that is not affected by pancreatic disease. To date, the investigators have validated their MRCP technique and have successfully performed both MR-PFT and MRE in CP patients; however normative data is essential for validation of our non-invasive technique.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between the ages of 6 and 15.9 years.
2. Subjects without a documented history of (or suggestive of) pancreatic disease

Exclusion Criteria:

1. History of pancreatic disease, liver disease, intra-abdominal neoplasm, abdominal inflammatory process such as inflammatory bowel disease (IBD), or systemic illness that may affect pancreatic state (e.g. cystic fibrosis).
2. Subjects with surgical hardware/implanted devices making them ineligible for MRI (e.g. pacemaker or other implanted medical device not approved for MRI).
3. Subjects who require any form of sedation or general anesthesia for MRI.
4. Subjects unable to breath-hold for the required 15-20 second imaging sequence.
5. Subjects who are pregnant or less than 12 months post-partum.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maisam Abu-El-Haija, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Andrew Trout, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amann ST, Yadav D, Barmada MM, O'Connell M, Kennard ED, Anderson M, Baillie J, Sherman S, Romagnuolo J, Hawes RH, Alkaade S, Brand RE, Lewis MD, Gardner TB, Gelrud A, Money ME, Banks PA, Slivka A, Whitcomb DC. Physical and mental quality of life in chronic pancreatitis: a case-control study from the North American Pancreatitis Study 2 cohort. Pancreas. 2013 Mar;42(2):293-300. doi: 10.1097/MPA.0b013e31826532e7. PMID 23357924
- [Background] Schwarzenberg SJ, Bellin M, Husain SZ, Ahuja M, Barth B, Davis H, Durie PR, Fishman DS, Freedman SD, Gariepy CE, Giefer MJ, Gonska T, Heyman MB, Himes R, Kumar S, Morinville VD, Lowe ME, Nuehring NE, Ooi CY, Pohl JF, Troendle D, Werlin SL, Wilschanski M, Yen E, Uc A. Pediatric chronic pancreatitis is associated with genetic risk factors and substantial disease burden. J Pediatr. 2015 Apr;166(4):890-896.e1. doi: 10.1016/j.jpeds.2014.11.019. Epub 2014 Dec 30. PMID 25556020
- [Background] Somaraju UR, Solis-Moya A. Pancreatic enzyme replacement therapy for people with cystic fibrosis. Cochrane Database Syst Rev. 2014 Oct 13;(10):CD008227. doi: 10.1002/14651858.CD008227.pub2. PMID 25310479
- [Background] Arya VB, Senniappan S, Demirbilek H, Alam S, Flanagan SE, Ellard S, Hussain K. Pancreatic endocrine and exocrine function in children following near-total pancreatectomy for diffuse congenital hyperinsulinism. PLoS One. 2014 May 19;9(5):e98054. doi: 10.1371/journal.pone.0098054. eCollection 2014. PMID 24840042
- [Background] Conwell DL, Zuccaro G Jr, Vargo JJ, Morrow JB, Obuchowski N, Dumot JA, Trolli PA, Burton A, O'laughlin C, Van Lente F. An endoscopic pancreatic function test with cholecystokinin-octapeptide for the diagnosis of chronic pancreatitis. Clin Gastroenterol Hepatol. 2003 May;1(3):189-94. doi: 10.1053/cgh.2003.50028. PMID 15017490
- [Background] Abu Dayyeh BK, Conwell D, Buttar NS, Kadilaya V, Hart PA, Baumann NA, Bick BL, Chari ST, Chowdhary S, Clain JE, Gleeson FC, Lee LS, Levy MJ, Pearson RK, Petersen BT, Rajan E, Steen H, Suleiman S, Banks PA, Vege SS, Topazian M. Pancreatic juice prostaglandin e2 concentrations are elevated in chronic pancreatitis and improve detection of early disease. Clin Transl Gastroenterol. 2015 Jan 29;6(1):e72. doi: 10.1038/ctg.2014.23. PMID 25630864
- [Background] Pelley JR, Gordon SR, Gardner TB. Abnormal duodenal [HCO3-] following secretin stimulation develops sooner than endocrine insufficiency in minimal change chronic pancreatitis. Pancreas. 2012 Apr;41(3):481-4. doi: 10.1097/MPA.0b013e31823a4c33. PMID 22228105
- [Background] Sendler M, Beyer G, Mahajan UM, Kauschke V, Maertin S, Schurmann C, Homuth G, Volker U, Volzke H, Halangk W, Wartmann T, Weiss FU, Hegyi P, Lerch MM, Mayerle J. Complement Component 5 Mediates Development of Fibrosis, via Activation of Stellate Cells, in 2 Mouse Models of Chronic Pancreatitis. Gastroenterology. 2015 Sep;149(3):765-76.e10. doi: 10.1053/j.gastro.2015.05.012. Epub 2015 May 19. PMID 26001927
- [Background] Conwell DL, Zuccaro G, Purich E, Fein S, Vanlente F, Vargo J, Dumot J, O'laughlin C, Trolli P. The effect of moderate sedation on exocrine pancreas function in normal healthy subjects: a prospective, randomized, cross-over trial using the synthetic porcine secretin stimulated Endoscopic Pancreatic Function Test (ePFT). Am J Gastroenterol. 2005 May;100(5):1161-6. doi: 10.1111/j.1572-0241.2005.41386.x. PMID 15842594
- [Background] Conwell DL, Zuccaro G, Purich E, Fein S, Vargo JJ, Dumot JA, VanLente F, Lopez R, Trolli P. Comparison of endoscopic ultrasound chronic pancreatitis criteria to the endoscopic secretin-stimulated pancreatic function test. Dig Dis Sci. 2007 May;52(5):1206-10. doi: 10.1007/s10620-006-9469-6. Epub 2007 Mar 27. PMID 17387611
- [Background] Zuccaro P, Stevens T, Repas K, Diamond R, Lopez R, Wu B, Conwell DL. Magnetic resonance cholangiopancreatography reports in the evaluation of chronic pancreatitis: a need for quality improvement. Pancreatology. 2009;9(6):764-9. doi: 10.1159/000201304. Epub 2010 Jan 21. PMID 20110743
- [Background] Sainani NI, Kadiyala V, Mortele K, Lee L, Suleiman S, Rosenblum J, Wang W, Banks PA, Conwell DL. Evaluation of Qualitative Magnetic Resonance Imaging Features for Diagnosis of Chronic Pancreatitis. Pancreas. 2015 Nov;44(8):1280-9. doi: 10.1097/MPA.0000000000000466. PMID 26465953
- [Background] Balci NC, Smith A, Momtahen AJ, Alkaade S, Fattahi R, Tariq S, Burton F. MRI and S-MRCP findings in patients with suspected chronic pancreatitis: correlation with endoscopic pancreatic function testing (ePFT). J Magn Reson Imaging. 2010 Mar;31(3):601-6. doi: 10.1002/jmri.22085. PMID 20187202
- [Background] Shi Y, Glaser KJ, Venkatesh SK, Ben-Abraham EI, Ehman RL. Feasibility of using 3D MR elastography to determine pancreatic stiffness in healthy volunteers. J Magn Reson Imaging. 2015 Feb;41(2):369-75. doi: 10.1002/jmri.24572. Epub 2014 Feb 5. PMID 24497052
- [Background] Itoh Y, Takehara Y, Kawase T, Terashima K, Ohkawa Y, Hirose Y, Koda A, Hyodo N, Ushio T, Hirai Y, Yoshizawa N, Yamashita S, Nasu H, Ohishi N, Sakahara H. Feasibility of magnetic resonance elastography for the pancreas at 3T. J Magn Reson Imaging. 2016 Feb;43(2):384-90. doi: 10.1002/jmri.24995. Epub 2015 Jul 7. PMID 26149267

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Participants: MRCP with Secretin and MR elastography will be performed on all participants.
  Secretin
Period: Overall Study
Arm/Group | Healthy Participants
Started | 57
Completed | 50
Not Completed | 7
Not completed — participant aversion to IV | 5
Not completed — participant fear of MRI scanner | 2

BASELINE CHARACTERISTICS:
Groups:
- Healthy Participants: Healthy participants will undergo Magnetic Resonance Imaging with secretin stimulation.
  Secretin
Arm/Group | Healthy Participants
Number analyzed (Participants) | 50
Age, Customized [Count of Participants; unit: Participants] — 50 participants
  Participants
    6-11 years | 27
    12-16 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 33
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Secreted Fluid Volume as Measured by MR-PFT
Description: Participants underwent MR imaging prior to and following secretin administration. Pre-secretin imaging lasts approximately 20 minutes. Post-secretin images were acquired at 1 minute, 5 minutes and 15 minutes following completion of secretin injection. Pre-secretin enteric fluid volumes were subtracted from post-secretin enteric fluid volumes for each participant to determine volume secreted in response to secretin administration at each time point.
  A commercially available software package determines the area of fluid signal on the MR images. The fluid signal from the pre-secretin images is then subtracted from the each post-secretin image (1, 5 and 15 minutes images) to determine the amount of fluid produced by the introduction of secretin.
Time Frame: 35 minutes (20 min pre-secretin, 15 minutes post-secretin)
Population: Healthy participants
Measure: Median (Full Range); unit: mL
Arm/Group | Healthy Participants
Number analyzed (Participants) | 50
mL | 79 [32 to 162]

2. Secondary Outcome: Pancreatic Stiffness as Measured by Magnetic Resonance Elastography (MRE)
Description: Healthy controls underwent 3D MRE on a 1.5T scanner. Regions of interest for measurement of pancreatic stiffness were drawn by two blinded readers and statistical analysis were performed for comparisons between the 2 groups.
Time Frame: Single time point, pre-secretin
Population: Of the 50 healthy controls recruited, complete MRE data were available for 49 subjects
Measure: Mean (Standard Deviation); unit: kPa
Groups:
- Healthy Participants: Healthy participants underwent MR elastography of the pancreas
Arm/Group | Healthy Participants
Number analyzed (Participants) | 49
kPa | 1.7 (0.3)

3. Secondary Outcome: Volumetric Measurement of Pancreatic Parenchymal Volume
Description: Pancreatic parenchymal volume by manual segmentation (tracing) of pancreas contours on magnetic resonance imaging (MRI)
Time Frame: Single time point, pre-secretin
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Healthy Participants
Number analyzed (Participants) | 50
mL | 46 (18.8)

ADVERSE EVENTS:
Time Frame: Approximately 2.5-3 hours
Description: Adverse events for this one visit study were collected from time of consent until completion of the study visit (approximately 2.5-3 hours)
Arm/Group | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 1/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants (N=50)
Nausea (Gastrointestinal disorders) | 1 (1) — No vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT02869893/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT02869893/ICF_001.pdf